CLINICAL TRIAL: NCT01899157
Title: Nutritional Status Among naïve HIV-infected Patients and HIV-infected Patients Receiving Highly Active Antiretroviral Therapy
Brief Title: Nutritional Status Among naïve HIV Infected Patients and HIV Infected Patients Receiving Highly Active Antiretroviral Therapy
Acronym: TNT-HIV 001
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: World Health Organization (Other); Bamrasnaradura Infectious Diseases Institute (Other Government); Ministry of Health, Thailand (Other Government); Mahidol University (Other); Chulalongkorn University (Other); BNH Hospital (Unknown)
Responsible Party: Principal Investigator, Nittaya Phanuphak, M.D., Dr., Thai Red Cross AIDS Research Centre
Other Study IDs: TNT-HIV001
Record Dates: First submitted 2013-06-06; First posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: Nutritional status; Nutritional situation
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey: 1. Thai naive HIV-infected patients
  2. Thai HIV-infected patient reciering highly active antiretroviral therapy

SUMMARY:
A prospective cross-sectional study evaluates nutritional status and its relationship to the related factors in Thai HIV-infected patients who attending in out patient clinic.

DETAILED DESCRIPTION:
A prospective cross-sectional study evaluates nutritional status and its relationship to the related factors in Thai HIV-infected patients who attending in out patient clinic at The Thai Red Cross AIDS Research Centre, Bamrasnaradura Infectious Disease Institute, Surat Thani hospital, Khonkaen hospital, Sanpathong hospital and the Queen Savang Vadhana Hospital at Sri Racha .

General Objective: To determine nutritional status among Thai People Living with HIV (PLHIV).

Specific Objective:

1. To assess nutritional problems including undernutrition, overnutrition and others such as lipodystrophy, dyslipidemia, hyperglycemia, cardiovascular disease, etc. among naïve HIV-infected patients and HIV-infected patients undergoing HARRT by using ABCDEF approach: Anthropometric, Biochemical, Clinical, Dietary, Exercise and Family assessment.
2. To describe the relationship between the nutritional status and HIV disease staging and other related factors among naïve HIV-infected patients and HIV-infected patients undergoing HARRT.
3. To describe the prevalence of CVD and its relationship to cardiac risk factors
4. To validate the community screening tool developed by the Thai Nutrition Taskforce in HIV (TNT-HIV) by assessing the correlation of this tool and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* 18 years of age or older
* Receiving ongoing care as part of the anonymous clinic, TRCARC, the antiretroviral therapy clinics at Bamrasnaradura Infectious Disease Institute, Surat Thani hospital, Khonkaen hospital, Sanpathong hospital and the Queen Savang Vadhana Hospital at Sri Racha.
* Either naïve HIV-infected patients and HIV-infected patients undergoing HARRT

Exclusion Criteria:

* HIV negative
* Patient who had active AIDS-related disorders within three months before participate the study
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 580 Thai HIV-infected patients who either did or did not receive treatment with antiretroviral therapy at The Thai Red Cross AIDS Research Centre, Bamrasnaradura Infectious Disease Institute, Surat Thani hospital, Khonkaen hospital, Sanpathong hospital and the Queen Savang Vadhana Hospital at Sri Racha.; These participants will be enrolled at TRCARC and Bamrasnaradura Infectious Disease Institute for amount 300 HIV infected patients and 70 HIV infected patients from each 4 region hospital.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Nutritional status and Nutritional situation | 1 year
  Nutritional status and Nutritional situation in Naïve HIV infected patients and HIV-infected patients undergoing HAART. It will be collected by using ABCDEF approch: Anthropometric, Biochemistry, Clinical, Dietary, Exercise and Family assesment.

SECONDARY OUTCOMES:
The prevalence of metabolic syndrome | 1 year
  The prevalence of metabolic syndrome in Naïve HIV infected patients and HIV-infected patients undergoing HARRT using American Heart Association (AHA) and National Heart Lung and Blood Institute (NHLBI) criteria

OTHER OUTCOMES:
The community screening tool | 1 year
  To validate the community screening tool developed by the Thai Nutrition Task Force for HIV (TNT-HIV) by assessing the correlation of this tool and nutritional status.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Wisit Prasithsirikul, Principal Investigator — Bamrasnaradura Infectious Disease Institute
Locations (1):
- Thai Red Cross AIDS Research Centre, Bangkok, Pathumwan, Thailand